CLINICAL TRIAL: NCT06410937
Title: Evaluation Of Drainless Thyroidectomy For Benign Thyroid Diseases Regarding Surgical Site Complications
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdelgaber Mehrez, resident of general surgery of sohag university, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Soh-Med-24-04-04MS
Record Dates: First submitted 2024-05-02; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Benign Thyroid Diseases
MeSH Terms: interventions — Thyroidectomy; Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drain used in the thyroid surgery (Active Comparator)
  Interventions: Procedure: thyroidectomy with drain
- No Drain used in the thyroid surgery (Active Comparator)
  Interventions: Procedure: thyroidectomy without drain

INTERVENTIONS:
Procedure: thyroidectomy without drain — thyroidectomy without subcutaneous suction drain
  Arms: No Drain used in the thyroid surgery
Procedure: thyroidectomy with drain — hyroidectomy with subcutaneous suction drain
  Arms: Drain used in the thyroid surgery

SUMMARY:
In all thyroid surgeries, many surgeons utilize drains on a regular basis and have done so for years according to recommendations. Due to the thyroid's high vascularization throughout its endocrine function, any haemorrhage inside the closed paratracheal space has the potential to impede venous and lymphatic drainage, which might result in airway blockage and laryngopharyngeal oedema. Surgeons routinely perform post-operative thyroid gland draining in the modern surgical field. The goal is to stop fluid from accumulating in the surgical wound site, which could constrict the patient's trachea and jeopardize their life.

Thyroid storm, hypocalcemia, hematoma/haemorrhage impairing airway, recurrent or superior laryngeal nerve damage, and wound problems such as wound infection are among the main post-operative consequences of thyroid surgery.

Some reports indicate the use of drains following thyroid surgery is not very beneficial. Some researchers have been prompted by this to consider whether drains should be inserted during thyroid surgery in which several research papers and meta-analyses have also failed to demonstrate the benefit of drainage in thyroid surgery. Blood clots in the drains could cause severe post-operative bleeding, preventing the surgeon from being notified. Difficult thyroidectomy cases might be predicted by factors linked to the patient, the thyroid, or the surgeon.

When thyroidectomies are performed under ideal conditions-that is, in a setting where good anatomical and physiological expertise is matched with meticulous surgical skills-complications are rare. The ability of the surgeon to do a thyroid surgery without difficulties is crucial. It is not possible to see routine drain use as a substitute for these components.

Percutaneous drains are frequently used in head and neck surgery cases. However, although effective at preventing post-operative haematoma formation, their use can also be associated with significant complications, including infection, fistulae, pain, psychosocial implications and most notably, prolongation of hospital stay.

Accordingly, some researchers that reject the use of intraoperative drains, there isn't a very high rate of wound hemorrhages following thyroid surgery. Additionally, other research indicates that there is no difference in the two groups' incidence of post-operative problems with and without drainage.

Nearly all surgeons utilize a closed vacuum drain after the intervention to avoid the deadliest complication, a smothering haemorrhage, which several studies suggest may not be essential

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years.
* Both sexes.
* Unilateral \ bilateral thyroid benign nodules, with preoperative fine-needle aspiration biopsy.

Exclusion Criteria:

* Surgical contraindications such as coagulation dysfunction.
* Retrosternal goiter.
* A history of cervical surgery.
* Sever Co-morbid diseases (uncontrolled diabetes, sever cardiopulmonary disease).
* Malignancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation Of Drainless Thyroidectomy For Benign Thyroid Diseases Regarding Surgical Site Complications | 6 months
  This study aims to compare the effectiveness of Drainless Versus Drainage after thyroidectomy operations regarding post-operative short-term surgical site complications as pain, infections, seroma, haematoma and gaping in patients with benign thyroid diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Prichard RS, Murphy R, Lowry A, McLaughlin R, Malone C, Kerin MJ. The routine use of post-operative drains in thyroid surgery: an outdated concept. Ir Med J. 2010 Jan;103(1):26-7. PMID 20222393
- [Background] Scerrino G, Paladino NC, Di Paola V, Morfino G, Amodio E, Gulotta G, Bonventre S. The use of haemostatic agents in thyroid surgery: efficacy and further advantages. Collagen-Fibrinogen-Thrombin Patch (CFTP) versus Cellulose Gauze. Ann Ital Chir. 2013 Sep-Oct;84(5):545-50. PMID 23502460
- [Background] Sakorafas GH. Historical evolution of thyroid surgery: from the ancient times to the dawn of the 21st century. World J Surg. 2010 Aug;34(8):1793-804. doi: 10.1007/s00268-010-0580-7. PMID 20401481
- [Background] Colak T, Akca T, Turkmenoglu O, Canbaz H, Ustunsoy B, Kanik A, Aydin S. Drainage after total thyroidectomy or lobectomy for benign thyroidal disorders. J Zhejiang Univ Sci B. 2008 Apr;9(4):319-23. doi: 10.1631/jzus.B0720257. PMID 18381807
- [Background] Morrissey AT, Chau J, Yunker WK, Mechor B, Seikaly H, Harris JR. Comparison of drain versus no drain thyroidectomy: randomized prospective clinical trial. J Otolaryngol Head Neck Surg. 2008 Feb;37(1):43-7. PMID 18479627